CLINICAL TRIAL: NCT04518865
Title: Treatment Effects of Herbst Appliance in Skeletal Class II Cases During Prepubertal and Postpubertal Periods: A Cone Beam Computed Tomographic Study
Brief Title: Treatment Effects of Herbst Appliance in Skeletal Class II Cases During Prepubertal and Postpubertal Periods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, khaled farouk, lecturer, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Herbst azhar
Record Dates: First submitted 2020-08-16; First posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Class II Malocclusion, Division 1
Keywords: Class II malocclusion.; prepubertal patients.; postpubertal patients.; Herbst appliance.
MeSH Terms: conditions — Malocclusion, Angle Class II; Overbite | interventions — Orthodontic Appliances, Functional

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pre-pubertal group. (Experimental): The patients were allocated into the pre-pubertal group based on their skeletal stage of maturation using the modified cervical vertebrae maturation Staging (CVMS) with skeletal maturity stages of CVMS II and CVMS III
  Interventions: Device: Herbst appliance
- post-pubertal group (Experimental): The patients were allocated into the post-pubertal group based on their skeletal stage of maturation using the modified cervical vertebrae maturation Staging (CVMS) with skeletal maturity stages of CVMS V and CVMS IV
  Interventions: Device: Herbst appliance

INTERVENTIONS:
Device: Herbst appliance — The bottom line of the study is to investigate the changes after Herbst appliance treatment and relate it to the pubertal status of the skeletal class II patients using CBCT.

SUMMARY:
The study was directed to compare the treatment outcomes of subjects with Class II malocclusion who were treated with Herbst appliance before and after puberty.

DETAILED DESCRIPTION:
Thirty-six Class II patients were randomly selected and divided into two groups based on their stage of skeletal maturation: pre-pubertal group (18 patients, mean age 9.15± 1.5 years) and post-pubertal group (18 patients, mean age 16.3 ± 1.0 years). All patients were treated with metallic splint supported Herbst IV appliance.

Pretreatment and post-Herbst IV treatment cone beam CT(CBCT) scans were obtained for both groups. Dentoskeletal and TMJ measurements made on the CBCT scans were analysed.

ELIGIBILITY:
Inclusion Criteria:

1. Skeletal Class II malocclusion with retrognathic mandible (ANB >5°, SNB<76°)
2. Normal growth pattern (SN/MP angle was in 25°- 35° range)
3. Unilateral or bilateral Class II molar relationship greater than or equal to one-half a cusp width.
4. Minimal or no crowding in the mandibular arch (0-5mm).
5. Average inclination or slight retroclination of the lower incisor.
6. An overjet greater than 5 mm.

Exclusion Criteria:

1. Skletal Class I
2. Craniofacial syndrome.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Skeletal and dental changes | 8 months
  The DICOM (Digital Imaging and Communications in Medicine) files from the pre and post CBCT scans were imported to Mimics software (Version 10.1, Materialise NV, Leuven, Belgium); and the cephalometric landmarks and planes were defined . Linear sagittal measurements of point A, point B, glenoid fossa, upper incisor, lower incisor, upper molars, and lower molars were recorded in relation to orbital perpendicular plane.

SECONDARY OUTCOMES:
Condylar head position | 8 months
  The Most middle-superior point of the mandibular condyle was determined in sagittal, axial and coronal views. In the sagittal slice of the middle condylar head, a line was drowned through the widest measurement of the condylar heads visible on the slice, from this line, three lines were raised crossing the glenoid fossa at 45°, 90°, and 135° . Four linear measurements representing the anterosuperior, superior, posterosuperior, and posterior distance were taken from the glenoid fossa wall to the surface of the condyle

CONTACTS AND LOCATIONS:
Overall Officials: khaled Farouk, lecturer, Principal Investigator — Al-Azhar University
Locations (1):
- Al-Azhar university, Cairo, Egypt